CLINICAL TRIAL: NCT01915641
Title: CPAP Improves the Walking Capacity in Patients With COPD and OSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 101-5303B
Record Dates: First submitted 2013-07-28; First posted 2013-08-05 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2013-04

CONDITIONS: Walking Capacity
Keywords: walking capacity; COPD; OSA; CPAP
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group A (Active Comparator): group A : CPAP treatment with optimal pressure for 1 month, repeat measurement change CPAP treatment to sham pressure 5cm H2O for 1 month, repeat measurement
  Interventions: Device: CPAP
- group B (Sham Comparator): group B : CPAP treatment with sham pressure for 1 month, repeat measurement change CPAP treatment with optimal pressure for 1 month, repeat measurement
  Interventions: Device: CPAP

INTERVENTIONS:
Device: CPAP — Randomized those patients to group A and group B group A : CPAP treatment with optimal pressure for 1 month, repeat measurement change CPAP treatment to sham pressure 5cm H2O for 1 month, repeat measurement group B : CPAP treatment with sham pressure for 1 month, repeat measurement change CPAP treatment with optimal pressure for 1 month, repeat measurement
  Other Names: continuous positive airway pressure

SUMMARY:
We have reported that CPAP treatment improved the walking capacity of overlap syndrome patients.

However, the previous study was not randomized, double blinded study. Therefore, we design a prospective, randomized, double blinded, controlled, cross-over trial to confirm this finding.

DETAILED DESCRIPTION:
inclusion criteria :

* COPD : FEV1/FVC < 70%, no response to bronchodilator (FEV1 change <12% and <200ml)
* OSA : AHI > 15/h, obstructive type predominant

exclusion criteria :

* any malignancy
* pregnancy
* claustrophobia
* age<18

primary outcome : exercise capacity (walking distance (meter), measured by incremental shuttle walking test)

Method : For those fit in criteria. CPAP titration will be performed to determine the optimal pressure Baseline measurement : incremental shuttle walking test, urine catecholamine, heart rate variability, muscle power and other baseline characteristics Randomized those patients to group A and group B group A : CPAP treatment with optimal pressure for 1 month, repeat measurement change CPAP treatment to sham pressure 5cm H2O for 1 month, repeat measurement group B : CPAP treatment with sham pressure for 1 month, repeat measurement change CPAP treatment with optimal pressure for 1 month, repeat measurement

ELIGIBILITY:
Inclusion Criteria:

* FEV1/FVC < 70%, no response to bronchodilator (FEV1 change <12% and <200ml)
* OSA : AHI > 15/h, obstructive type predominant

Exclusion Criteria:

* any malignancy
* pregnancy
* claustrophobia
* age<18

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-04; Primary Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
exercise capacity (walking distance (meter), measured by incremental shuttle walking test) | CPAP treatment for 1 month

CONTACTS AND LOCATIONS:
Overall Officials: TSAI-YU WANG, MD, Principal Investigator — Department of Thoracic Medicine, Chang Gung Memorial Hospital 199 Tun-Hwa N. Rd., Taipei, Taiwan; TSAI-YU WANG, MD, Principal Investigator — Department of Thoracic Medicine, Chang Gung Memorial Hospital
Locations (1):
- Department of Thoracic Medicine, Chang Gung Memorial Hospital, Taipei, Taiwan